

September 04, 2020 



## **PROTOCOL #16-308**

**XIENCE 90 Study** 

**Statistical Analysis Plan** 

**September 04, 2020** 

# **Confidential and Proprietary**

Nothing herein is to be disclosed without the expressed written consent of Abbott Vascular

#### TABLE OF CONTENTS



| 1. S | YNOPSIS OF STUDY DESIGN AND PROCEDURES | 4 |
|---|---|---|
| 1.1 | Purpose of the Statistical Analysis Plan | 4 |
| 1.2 | Study Objectives | 4 |
| 1.3 | Study Design | 4 |
| | 1.3.1 Selection of Control | 5 |
| | 1.3.2 Primary Endpoint | 6 |
| | 1.3.3 Secondary Endpoint(s) | 6 |
| | 1.3.3.1 Major Secondary Endpoint(s) | 6 |
| | 1.3.3.2 Other Secondary Endpoint(s) | 6 |
| 1.4 | Analysis Populations | 7 |
| | Primary Analysis Population | 7 |
| 1.5 | Sample Size Calculations | |
| | | 8 |
| | | 8 |
| | | 9 |
| 2. A | NALYSIS CONSIDERATIONS | 10 |
| 2.1 | Statistical Methods | 10 |
| | 2.1.1 Descriptive Statistics for Continuous Variables | 10 |
| | 2.1.2 Descriptive Statistics for Categorical Variables | 12 |
| | 2.1.3 Propensity Score | |
| | 2.1.3-1 Propensity Score Variable List | 15 |
| | 2.1.4 Hypothesis Testing | |
| | I. Major Secondary Endpoint #1: Bleeding rate (BARC type 2-5) from 3- to 12-month fo | ollow- |
| | up 18 | |
| | II. Major Secondary Endpoint #2: Stent Thrombosis (ARC definite/probable) from 3- to 1 | 12- |
| | month follow-up | 18 |
| | 2.1.5 Survival Analyses | 19 |
| 2.2 | Endpoint Analyses | 19 |
| | 2.2.1 Primary Endpoint Analysis | 19 |
| | 2.2.2 Major Secondary Endpoint Analysis | 19 |
| | 2.2.3 Secondary Endpoint Analyses | |
| 2.3 | Subgroups for Analysis | 20 |
| | 2.3.1 Sex | 20 |
| | 2.3.2 Diabetes | 20 |
| | 2.3.3 Covid-19 pandemic impact | 20 |
| | 2.3.4 Other Subgroups | 20 |
| 2.4 | Analysis Window | |
| 2.5 | Handling of Missing Data | |
| 2.6 | Poolability Issue | |
| | 2.6.1 Multiple Geography Effect | |
| | 2.6.2 Multiple Center Effect | |
| 2.7 | Adjustments for Covariates | |
| 2.8 | Multiplicity Issues | |
| 2.0 | Muliphely issues | ∠∠ |



September 04, 2020 

| 2.10 Documentation and Other Considerations | 24 |
|---------------------------------------------|----|
| 3. ACRONYMS AND ABBREVIATIONS | 25 |
| 4. REFERENCES | |



September 04, 2020 

#### 1. SYNOPSIS OF STUDY DESIGN AND PROCEDURES

#### 1.1 **Purpose of the Statistical Analysis Plan**

This statistical analysis plan (SAP) is intended to provide a detailed and comprehensive description of the planned methodology and analysis to be used for Protocol 16-308 the XIENCE May 25, 2018 study protocol. 90 clinical study. This plan is based on the

#### 1.2 **Study Objectives**

**Primary Objective:** to show non-inferiority of the primary endpoint of all death or all MI (modified ARC) from 3 to 12 months following XIENCE implantation in HBR subjects treated with 3-month DAPT compared to a historical control after propensity score adjustment.

#### **Secondary Objective:**

- To show superiority of the major secondary endpoint of major bleeding (Bleeding Academic Research Consortium [BARC] type 2-5) from 3 to 12 months following XIENCE implantation in HBR subjects treated with 3-month DAPT compared to a historical control after propensity score adjustment.
- To evaluate stent thrombosis (ARC definite/probable) from 3 to 12 months following XIENCE implantation in HBR subjects treated with 3-month DAPT against a performance goal (PG).

#### 1.3 **Study Design**

XIENCE 90 study is a prospective, single arm, multi-center, open label trial to evaluate the safety of 3-month dual antiplatelet therapy (DAPT) in subjects at high risk of bleeding (HBR) undergoing percutaneous coronary intervention (PCI) with the approved XIENCE family of coronary drug-eluting stents.

The XIENCE family stent systems include commercially approved XIENCE Xpedition Everolimus Eluting Coronary Stent System (EECSS), XIENCE Alpine EECSS or XIENCE PROX EECSS (OUS only)<sup>b</sup>, XIENCE PROA EECSS (OUS only)<sup>c</sup>, and XIENCE Sierra EECSS,

<sup>&</sup>lt;sup>a</sup> The commercially approved XIENCE stent will be used in geographies where it is commercially available

<sup>&</sup>lt;sup>b</sup> XIENCE PRO<sup>X</sup> is a rebrand of the XIENCE Xpedition Stent System and is only available outside of the United

<sup>&</sup>lt;sup>c</sup> XIENCE PRO<sup>A</sup> is a rebrand of the XIENCE Alpine Stent System and is only available outside of the United States.

September 04, 2020 

which are all manufactured by Abbott Vascular, Inc, Santa Clara, USA. The above XIENCE family stent systems will hereinafter be called "XIENCE" in this study.

Approximately 2,000 subjects from approximately 100 sites globally will be registered in this study, with at least 50% of subjects in the United States (US). Study population consists of noncomplex HBR subjects with up to three native coronary artery lesions (a maximum of two lesions per epicardial vessel) with reference vessel diameter between 2.25 mm and 4.25 mm. Eligibility of P2Y12 receptor inhibitor discontinuation will be assessed at 3-month follow-up. Subjects who are free from myocardial infarction (modified ARC), repeat coronary revascularization, stroke, or stent thrombosis (ARC definite/probable) within 3 months (prior to 3-month visit but at least 90 days) after stenting AND have been compliant with 3-month DAPT without interruption of either aspirin and/or P2Y12 receptor inhibitor for > 7 consecutive days are considered as "3-month clear", and will discontinue P2Y12 receptor inhibitor and continued with aspirin monotherapy after 3-month follow-up.

All registered subjects will be followed at 3, 6 and 12 months post index procedure.

The data collected from the XIENCE 90 study will be compared with the historical control of non-complex HBR subjects treated with standard DAPT duration of up to 12 months from the XIENCE V USA study, which is a US post-approval study to evaluate the safety of XIENCE V EECSS in "all-comer" population under real-world setting.

#### 1.3.1 Selection of Control

The XIENCE V USA historical HBR control for 3-month DAPT study is derived based on the following criteria:

## **Definition of non-complex HBR from XIENCE V USA**

- HBR inclusion criteria (any one of the below HBR criteria):
  - Age  $\geq$  75 years
  - History of major bleeding
  - History of stroke
  - o Receiving or scheduled to receive chronic anticoagulation therapy
  - o Renal insufficiency (creatinine > 2mg/dl)
  - Anemia (Hb < 11g/dl or transfusion)
  - o Thrombocytopenia (platelet count < 100.000/mm3)
- Exclusion criteria for non-complex:
  - o STEMI
  - o LVEF < 30%
  - o Patients with more than 3 lesions treated during index procedure
  - o Patients with more than 2 vessels treated during index procedure

September 04, 2020 

- $\circ$  At least one lesion with RVD < 2.25 mm or > 4.25 mm (visual estimation)
- At least one lesion located in left main
- o At least one lesion located in graft
- o At least one in-stent restenosis lesion
- At least one lesion containing thrombus
- o At least one target lesion having TIMI flow 0
- At least one target lesion with length > 32 mm by visual estimation.

The above selection criteria for the XIENCE V USA historical control aligns with the key inclusion/exclusion criteria of the XIENCE 90 Study.

For primary analysis, the XIENCE V USA non-complex HBR control subjects must be also 3-month clear, following the same logic as defined for the primary analysis population (refer to Section 1.4).

#### 1.3.2 Primary Endpoint

The primary endpoint is a composite rate of all death or all myocardial infarction (Academic Research Consortium [ARC]) from 3 months to 12 months.

#### 1.3.3 Secondary Endpoint(s)

#### 1.3.3.1 Major Secondary Endpoint(s)

- Major bleeding rate (BARC type 2-5) from 3 to 12 months.
- Stent thrombosis (ARC definite/probable) from 3 to 12 months

#### 1.3.3.2 Other Secondary Endpoint(s)

The following endpoints will be assessed from 3 to 12 months:

- All death, cardiac death, vascular death, non-cardiovascular death
- All MI (modified ARC) and MI attributed to target vessel (TV-MI, modified ARC)
- Composite of cardiac death or MI (modified ARC)
- All stroke, ischemic stroke and hemorrhagic stroke
- Clinically-indicated target lesion revascularization (CI-TLR)
- Clinically-indicated target vessel revascularization (CI-TVR)
- Target lesion failure (TLF, composite of cardiac death, TV-MI and CI-TLR)
- Target vessel failure (TVF, composite of cardiac death, TV-MI and CI-TVR)
- Major bleeding defined by the Bleeding Academic Research Consortium (BARC) type 3-

September 04, 2020 

# 1.4 Analysis Populations

# **Primary Analysis Population**

| The primary analysis population includes "3-month clear" population, defined as subjects who are free from myocardial infarction (modified ARC), repeat coronary revascularization, stroke, or stent thrombosis (ARC definite/probable) within 3 months after stenting AND have been compliant with 3-month dual antiplatelet therapy (DAPT) |
|---|
| • |
| 1.5 Sample Size Calculations |
| <ul> <li>Sample size in the control arm (3-month clear): ~1,150</li> </ul> |
| A total sample size of 2,000 subjects in the XIENCE 90 study will be required for this test. |









September 04, 2020 





#### 2. ANALYSIS CONSIDERATIONS

#### 2.1 Statistical Methods

Baseline demographic, clinical, angiographic, procedural, and device data, and clinical results will be summarized using descriptive summary statistics.

#### **Descriptive Statistics for Continuous Variables** 2.1.1

For continuous variables (e.g., age, percent diameter stenosis and lesion length), results will be summarized with the numbers of observations, means, and standard deviations and where specified in the table mockups, with quartiles, minimums, maximums, and two-sided 95% confidence intervals for the means as per the table mockups. Differences between two comparison groups of interest, where specified, will be summarized with the differences of the two means, and two-sided 95% confidence intervals for the difference between the means. These calculations will be done under the assumption that the data for the two arms are independent and approximately normal in distribution. The confidence interval for the difference of two means will be calculated under the assumption of unequal variances. If the asymptotic assumptions fail, then nonparametric summary statistics (medians, 25th and 75th percentiles) may be displayed as an alternative.

Formulas for calculation of the confidence intervals for the continuous variables are given below:

1. 100(1- α)% Confidence Interval For A Single Mean<sup>5</sup>

$$\bar{x} \pm t_{\frac{\alpha}{2}} \frac{s}{\sqrt{n}}$$

where:

 $\bar{x}$  = sample mean

s = sample standard deviation

n = sample size

 $t_{\underline{\alpha}}$  = the alpha/2 t - statistic for n-1 degrees of freedom

2. 100(1-α)% Confidence Interval For The Difference of Two Means Under The Assumption Of Equal Variances Between The Two Groups<sup>5</sup>

$$(\overline{x}_1 - \overline{x}_2) \pm t_{\frac{\alpha}{2}} \sqrt{s_p^2 \left(\frac{1}{n_1} + \frac{1}{n_2}\right)}$$

September 04, 2020 

where:

$$\bar{x}_1$$
 = sample mean for group 1

 $\overline{x}_2$  = sample mean for group 2

$$s_p^2 = \frac{(n_1 - 1)s_1^2 + (n_2 - 1)s_2^2}{n_1 + n_2 - 2}$$

 $s_1$  = sample standard deviation for group 1

 $s_2$  = sample standard deviation for group 2

$$n_1$$
 = sample size for group 1

 $n_2$  = sample size for group 2

$$t_{\frac{\alpha}{2}}$$
 = the alpha/2 t - statistic for  $n_1 + n_2 - 2$  degrees of freedom

3. 100(1-α) % Confidence Interval for the Difference of Two Means under the Assumption of Unequal Variances between the Two Groups<sup>5</sup>

$$(\overline{x}_1 - \overline{x}_2) \pm t_{\frac{\alpha}{2}} SED$$

With the degrees of freedom for the approximate t statistic is determined by Satterthwaite's formula<sup>2</sup> as follows:

$$df = \frac{\left(w_1 + w_2\right)^2}{\frac{w_1^2}{n_1 - 1} + \frac{w_2^2}{n_2 - 1}}$$

where:

 $\bar{x}_1$  = sample mean for group 1

 $\overline{x}_2$  = sample mean for group 2

 $s_1$  = sample standard deviation for group 1

 $s_2$  = sample standard deviation for group 2

 $n_1 =$ sample size for group 1

 $n_2$  = sample size for group 2

$$SED = \sqrt{\frac{{s_1}^2}{n_1} + \frac{{s_2}^2}{n_2}}$$

$$w_1 = \frac{{s_1}^2}{n_1}$$




$$w_2 = \frac{{s_2}^2}{n_2}$$

#### 2.1.2 Descriptive Statistics for Categorical Variables

For categorical variables such as gender, Death/MI and TLF, results will be summarized with subject counts and percentages/rates, with exact two-sided 95% Clopper-Pearson<sup>6</sup> confidence intervals. Differences between two comparison groups of interest, when specified, will be summarized with the difference in percentages and the Newcombe<sup>5</sup> score two-sided 95% confidence interval for the difference of two percentages.

For efficacy and safety endpoint(s), relative risks (i.e., the ratio of rates), confidence interval for the relative risks, the difference in rates and the confidence interval for difference in rates (using previously-described formulas), and p-values may also be presented for hypothesis generating purposes. The p-values will be based on either Pearson's Chi-square test or Fisher's exact test by checking the expected frequency for each cell in the 2x2 contingency table against Cochran's rule<sup>8</sup>, i.e., if the expected frequencies for all cells are  $\geq 5$ , then Pearson's Chi-square test will be used, otherwise Fisher's exact test will be used.



Formulas for calculating confidence intervals for the categorical variables are given below.

1. 100(1-α) % Exact Clopper-Pearson Confidence Interval for A Single Proportion<sup>6</sup>

September 04, 2020 

Lower Confidence Limit = 
$$\frac{x}{x + (n - x + 1)F_{1 - \frac{\alpha}{2}}(2(n - x + 1), 2x)}$$

Upper Confidence Limit = 
$$\frac{(x+1)F_{1-\frac{\alpha}{2}}(2(x+1),2(n-x))}{n-x+(x+1)F_{1-\frac{\alpha}{2}}(2(x+1),2(n-x))}$$

where:

n =sample size

x = number of "events"

$$F_{1-\frac{\alpha}{2}}(df_1,df_2)$$
 = the (1-alpha/2) F-statistic for degrees of freedom  $df_1$  and  $df_2$ 

- 2. 100(1-α) % Newcombe Score Confidence Interval for the Difference of Two Proportions <sup>7</sup>
  - a. 100(1-α) % Wilson Score Confidence Interval for A Single Proportion<sup>5</sup>

Lower Confidence Limit = 
$$\left(\hat{p} + Z_{\alpha/2}^2 / 2n - Z_{\alpha/2} \sqrt{\left(\hat{p}(1-\hat{p}) + Z_{\alpha/2}^2 / 4n\right)/n}\right) / \left(1 + Z_{\alpha/2}^2 / n\right)$$

Upper Confidence Limit =  $(\hat{p} + Z_{\alpha/2}^2 / 2n + Z_{\alpha/2} \sqrt{(\hat{p}(1-\hat{p}) + Z_{\alpha/2}^2 / 4n)/n})/(1 + Z_{\alpha/2}^2 / n)$ where:

$$\hat{p} = x / n$$

n = sample size

x = number of "events"

 $Z_{\alpha/2} = 100(1 - \alpha/2)$ th percentile of the standard normal distribution

b. 100(1-α) % Newcombe Score Confidence Interval for the Difference of Two Proportions<sup>4</sup>



Lower Confidence Limit = 
$$(\hat{p}_1 - \hat{p}_2) - Z_{\alpha/2} \sqrt{L_1(1-L_1)/n_1 + U_2(1-U_2)/n_2}$$
  
Upper Confidence Limit =  $(\hat{p}_1 - \hat{p}_2) + Z_{\alpha/2} \sqrt{U_1(1-U_1)/n_1 + L_2(1-L_2)/n_2}$   
where:

 $\hat{p}_1 = \text{sample proportion for group 1}$ 

 $\hat{p}_2$  = sample proportion for group 2

 $L_1$  and  $U_1$  are the lower and upper Wilson Score confidence limits for  $p_1$   $L_2$  and  $U_2$  are the lower and upper Wilson Score confidence limits for  $p_2$ 

 $Z_{\alpha/2} = 100(1 - \alpha/2)$ th percentile of the standard normal distribution

#### 2.1.3 Propensity Score

Given that subjects in the two comparison groups (XIENCE 90 vs XIENCE V USA) are not randomized and thus may not have balanced baseline characteristics, the non-inferiority and superiority tests for 3-12 month period will be carried out through stratified analysis in the "3-month clear" population. The stratification will be performed through propensity scores (PS). For each individual a propensity score (i.e., predicted probability between 0 and 1) for group (XIENCE 90) membership will be calculated using logistics regression, with "group" as the outcome and baseline variables including demographic, lesion characteristics, and risk factors as the predictors. Subjects will be categorized into 5 groups based on the calculated propensity scores and their quintiles. Non-inferiority and superiority will then be carried out for the rate of the endpoint using the method described in sections below stratified by the propensity quintiles.

The propensity score modeling and design will be performed by an independent statistician who has no access to any outcome data of both the XIENCE 90 study and the XV USA historical control for the integrity and interpretability of study results. The independent statistician will be blinded and have no access to clinical outcome and any follow-up information to avoid introducing bias into the analysis.

September 04, 2020 



Per the recent publication by Yue et al<sup>28</sup> on two-stage study designs involving propensity score adjustment, the propensity score calculation results will subsequently be sent to the FDA for review and approval prior to performing the primary endpoint and major secondary endpoint analyses.

## 2.1.3-1 Propensity Score Variable List

Based on prior clinical experience and clinical research, below is the list of variables that are considered to be related to assignments modeling building:

- Gender
- Age
- Creatinine
- Chronic anticoagulant
- History of stroke
- History of major bleeding
- Platelet
- Hb
- BMI
- Hypertension
- Dyslipidemia
- Prior PCI
- Prior CABG

September 04, 2020 

- Prior MI
- Multivessel disease
- Clinical Presentation (ACS (NSTEMI, ACS unstable angina) vs. non-ACS)
- Diabetes
- ACC/AHA lesion complexity
- Total lesion length per patient
- RVD
- Diameter stenosis%
- Bifurcation
- Number of lesions treated
- Number of vessel treated
- Number of stents per patient
- Total stent length per patient
- Discharge P2Y12
- Paris bleeding score
- PRECISE DAPT score

## 2.1.4 Hypothesis Testing

#### Primary endpoint analysis for 3-month DAPT

The XIENCE 90 study is powered based on primary endpoint of Death/MI between 3-month and 12-month follow-up. Death/MI is defined as the composite endpoint of all death or all myocardial infarction (Academic Research Consortium [ARC]). This primary endpoint will be evaluated between XIENCE 90 and XIENCE V USA historical control stratified by propensity score quintiles in the primary analysis population.

The stratified Farrington-Manning method will be performed to test non-inferiority (NI) of 3month DAPT from XIENCE 90 compared to standard DAPT duration up to 12 months from




Abbott

XIENCE V USA historical control.



$$\hat{\delta}_{i} = p_{it} - p_{ic}$$

$$w_{i} = \frac{(N_{it} + N_{ic})}{\sum_{i} (N_{it} + N_{ic})}$$

$$V(\hat{\delta}_{i}) = \frac{p_{imt} (1 - p_{imt})}{N_{it}} + \frac{p_{imc} (1 - p_{imc})}{N_{ic}}$$

 $P_{imt}$  and  $P_{imc}$  are calculated as follows:

$$\begin{array}{l} r_i = N_{it}/N_{ic} \\ a1 = -\left(\ 1 + r_i + p_{ic} + r_i\ *p_{it} - \delta\ *(\ r_i + 2)\ \right) \\ a2 = \delta\ **2 - \delta\ *(2*p_{ic} + r_i + 1) + p_{ic} + r_i\ *p_{it} \\ a3 = p_{ic}\ *\delta\ *(1 - \delta) \\ u = a1**3/(3 + 3*\ r_i)**3 - a1*a2/(6*(1 + r_i)**2) + a3/(2 + 2*\ r_i) \\ v = sign(u)*sqrt(\ a1**2/((3 + 3*\ r_i)^**2) - a2/(3 + 3*\ r_i)) \\ w = 1/3*(\ arcos(-1) + arcos(u/v**3)) \\ p_{imc} = 2*v*cos(w) - a1/(3 + 3*\ r_i) \\ p_{imt} = p_{imc} + \delta \end{array}$$

#### Major secondary endpoints analyses for 3-month DAPT

If the hypothesis testing for the primary endpoint is successful, the hypotheses testing for the major secondary endpoint #1 will be performed followed by the hypotheses test for the major secondary endpoint #2.



September 04, 2020 

# I. Major Secondary Endpoint #1: Bleeding rate (BARC type 2-5) from 3- to 12-month follow-up

| The superiority test for the major secondary endpoint #1 will be performed stratified by |
|---|
| propensity score quintiles in the primary analysis population. |
| II. Major Secondary Endpoint #2: Stent Thrombosis (ARC definite/probable) from 3- to |
| 12-month follow-up |
| The exact test will be performed for major secondary endpoint #2 in the primary analysis |
| population. |

September 04, 2020 

This test will be performed if the superiority of major secondary endpoint #1 is established.

#### 2.1.5 Survival Analyses

Survival analysis may be conducted to analyze time-to-event variables. Subjects without events will be censored at their last known event-free time point. Survival curves will be constructed using Kaplan-Meier estimates.

Summary tables for the endpoints will include failure rates (Kaplan-Meier estimates). For the primary analysis report, all available data will be used.

#### 2.2 Endpoint Analyses

## 2.2.1 Primary Endpoint Analysis

#### **Primary Analysis:**

A non-inferiority test will be performed on the primary endpoint for the primary analysis population of the XIENCE 90 study and the XIENCE V USA historical control stratified by propensity score quintiles

To ensure all subjects to be included in this analysis, multiple imputations will be performed in calculating the propensity scores.

#### Secondary Analysis (as a sensitivity analysis):

In addition to the primary analysis stratified by propensity score quintile, a non-inferiority test will be performed on the primary endpoint stratified by propensity score quartile, with the same methodology as described above.

#### 2.2.2 Major Secondary Endpoint Analysis

The stratified Farrington and Manning method will be used for the stratified superiority test of major secondary endpoint #1 between 3-month and 12-month follow up for the primary analysis population of XIENCE 90 and XIENCE V USA historical control. The stratification is performed by propensity score quintiles.

To ensure all subjects to be included in this analysis, multiple imputations will be performed in calculating the propensity scores.

The exact test will be used for stent thrombosis between 3-month and 12-month follow-up against a PG for the primary analysis population as described in section 2.1.4. This test will be performed if the superiority of major secondary endpoint #1 is established.

#### 2.2.3 Secondary Endpoint Analyses

Other secondary clinical endpoints will be descriptively analyzed for both the primary analysis population and all registered subjects without propensity stratification.

#### 2.3 Subgroups for Analysis

All of the following subgroup analyses are intended for the primary analysis population. The comparison between the XIENCE 90 study and the XIENCE V USA historical control will analyzed descriptively within each quintile for the primary and major secondary endpoints in a specific subgroup. The above quintiles are based on the overall PS, not PS built within each subgroup, as baseline characteristics of subjects are likely to be comparable in each quintile of the overall PS.

#### 2.3.1 Sex

Sex-specific subgroup analyses will be performed on primary analysis population for the primary endpoint and the major secondary endpoints stratified by the overall PS.

#### 2.3.2 Diabetes

Diabetic subgroup analysis will be performed on primary analysis population for the primary and major secondary endpoints stratified by the overall PS. Analyses will be performed within the following subgroups:

- All diabetes mellitus, defined as any diabetics with or without medical treatment
- Non diabetes mellitus.

## 2.3.3 Covid-19 pandemic impact

In order to assess the COVID-19 impact on the primary endpoint and major secondary endpoints, a descriptive subgroup comparison will be performed on the primary analysis population between subjects whose primary endpoint follow-up overlaps with the pandemic outbreak (such as March 01, 2020 and after) and those whose primary endpoint follow-up is prior to the pandemic outbreak.

#### 2.3.4 Other Subgroups

The following subgroups will be evaluated for the primary analysis population for the primary and major secondary endpoints stratified by the overall PS. Analyses will be performed within the following subgroups:

September 04, 2020 

- Ethnicity (white versus non-white)
- Age (age  $\geq$  median vs < median)
- Age  $\geq$  65 years old (US elderly patient)
- Clinical presentation (ACS NSTEMI, ACS unstable angina, non-ACS)

#### 2.4 Analysis Window

- 6 months
- 12 months

# 2.5 Handling of Missing Data

The primary and major secondary endpoint analyses will be evaluated after propensity score stratification. To handle missing data in propensity score building, multiple imputation method will be performed for baseline characteristics to compute propensity scores from these datasets.

All other analyses will be based on available data with missing data excluded. Any unused or spurious data will be noted as appropriate in the final report.

## 2.6 Poolability Issue

#### 2.6.1 Multiple Geography Effect

Analysis will be performed by pooling data between geographies (US and OUS). XIENCE 90 study will enroll 2,000 subjects from approximately 100 sites globally, with at least 50% of subjects in the United States (US).

To evaluate the geography effect on the primary endpoint, Fisher's exact test will be tested for geography effect in the XIENCE 90 study against an alpha level of 0.05.

If the p-value is < 0.05, Abbott Vascular will examine subject demographics, baseline clinical, and angiographic characteristics for possible correlations and confounding factors.

#### 2.6.2 Multiple Center Effect

Analysis will be performed by pooling data across study sites.

The XIENCE 90 study will have 100 sites globally, with at least 50% of subjects in the United States. Subject registration is capped at 300 per site. This cap per site will prevent the scenario



where the results from a few sites dominate the overall study result. For the analysis of center effect, data from smaller sites may be combined for the analysis. Smaller sites are defined as sites with fewer than 20 subjects per site.



# 2.7 Adjustments for Covariates

Unless otherwise specified, no adjustments for covariates will be made for any of the variables in the analyses.

# 2.8 Multiplicity Issues

No multiplicity adjustment is necessary because the tests in this analysis plan are sequential.



## 2.9 Sensitivity Analysis

The primary and major secondary endpoints between 3-month and 12-month follow-up will be analyzed descriptively for the 3-month clear population removing the patients who do not have antiplatelet medication compliance after 3 months.

For the 3-month DAPT arm, antiplatelet medication non-compliance beyond 3-month follow-up for 3-month clear population is defined as patients who resume P2Y12 inhibitor for more than 7 consecutive days, and/or interrupt aspirin for more than 7 consecutive days between 3-month and 12-month follow up.



In addition, a sensitivity analysis will be performed for the primary endpoint analysis to evaluate the impact of the missing outcome. The analysis will be carried out based on the primary analysis population, and by imputing the missing outcomes for each imputed baseline PS dataset, and Rubin's combination rule [29] will be used to consolidate the final analysis for the 10 duplicates of the imputed dataset. Refer to Appendix A for more details.

September 04, 2020 

## 2.10 Documentation and Other Considerations

All analyses will be performed using SAS® for Windows, version 9.1 or higher.

September 04, 2020 

## 3. ACRONYMS AND ABBREVIATIONS

| Acronym or Abbreviation | Complete Phrase or Definition |
|-------------------------|-------------------------------------------------|
| ACS | Acute Coronary Syndrome |
| AMI | Acute Myocardial Infarction |
| ARC | Academic Research Consortium |
| BARC | Bleeding Academic Research Consortium |
| BMI | Body Mass Index |
| CABG | Coronary artery bypass grafting |
| CTO | Chronic Total Occlusion |
| DAPT | Dual Antiplatelet Therapy |
| DMR | Death/MI/Revascularization |
| EECSS | <b>Everolimus Eluting Coronary Stent System</b> |
| Hb | Hemoglobin |
| HBR | High Bleeding Risk |
| LVEF | Left Ventricular Ejection Fraction |
| MI | Myocardial Infarction |
| NSTEMI | non ST-segment elevation MI |
| PCI | Percutaneous Coronary Syndrome |
| PS | Propensity Score |
| RVD | Reference Vessel Diameter |
| SAP | Statistical Analysis Plan |
| ST | Stent Thrombosis |
| STEMI | ST-segment elevation myocardial infarction |
| TLF | Target Lesion Failure |
| TLR | Target Lesion Revascularization |
| TVR | Target Vessel Revascularization |
| US | United State |

September 04, 2020 

#### 4. REFERENCES

- 1. Li, H., Mukhi, V., Lu, N., Xu, Y.L. and Yue, L.Q., 2016. A Note on Good Practice of Objective Propensity Score Design for Premarket Nonrandomized Medical Device Studies with an Example. *Statistics in Biopharmaceutical Research*, 8(3), pp.282-286.
- 2. D'Agostino, R.B., 1998. Tutorial in biostatistics: propensity score methods for bias reduction in the comparison of a treatment to a non-randomized control group. *Stat Med*, 17(19), pp.2265-2281.
- 3. Farrington, C. P., Manning, G., Test Statistics and Sample Size Formulae for Comparative Binomial Trials with Null Hypothesis of Non-Zero Risk Difference or Non-Unity Relative Risk. Statistics in Medicine, 1990, 9, 1447-1454.
- 4. Hintze J. NCSS and PASS. Number Cruncher Statistical Systems. Kaysville, Utah. 2005.
- 5. SAS/STAT® 9.2 User's Guide, Second Edition, SAS Institute Inc., Cary, NC, 2009.
- 6. Clopper C. J., Pearson E. S., The Use of the Confidence or Fiducial Limits Illustrated in the Case of the Binomial. Biometrika, 1934, 26, 404-413.
- 7. Newcombe, R. G., Interval estimation for the difference between independent proportions: comparison of eleven methods, Statistics in Medicine, 1998, 17, 873-890.
- 8. Cochran, W. G., Some Methods for Strengthening the Common  $\chi^2$  Test. Biometrics, 1954, 10, 417-451.
- 9. Wilson, E. B., Probable inference, the law of succession, and statistical inference, Journal of the American Statistical Association, 1927, 22, 209-212.
- 10. Draft Guidance for Industry and Food and Drug Administration Staff: Evaluation of Sex Differences in Medical Device Clinical Studies, December 19, 2011, CDRH
- 11. Gail, M., Simon, R., Testing for Qualitative Interactions between Treatment Effects and Patient Subsets, Biometrics, 1985, 41, 361-372.
- 12. Dmitrienko, A. et. al., Analysis of Clinical Trials Using SAS: A Practical Guide, SAS Institute, Cary, NC, 2005.
- 13. Fleming TR& Harrington DP 1991. Counting Processes and Survival Analysis. New York: Wiley.
- 14. Miller R & Halpern J 1982. Regression with censored data. Biometrika 69, 521-31.
- 15. Allison PD. Survival Analysis Using the SAS system: A Practical Guide, Cary, NC: SAS Institute Inc., 1995.
- 16. Kaplan EL, Meier P. Non-parametric estimation from incomplete observations. J Am Stat Assoc 1958; 53:457-481.
- 17. Therneau TM, Grambsch PM. Modeling survival data: extending the Cox model. New York: Springer-Verlag; 2000.
- 18. Allison PD. Multiple Imputation for Missing Data. Sociological Methods & Research, Feb 2000; Vol. 28 No. 3:301-309.

September 04, 2020 

- 19. Barnes SA, Lindborg SR, Seaman JW. Multiple Imputation Techniques in Small Sample Clinical Trials. Stat Med 2006 Jan 30; 25(2):233-45.
- 20. Clopper CJ, Pearson E. The Use of the Confidence or Fiducial Limits Illustrated in the Case of the Binomial. Biometrika 1934; 26:404-413.
- 21. Lavori PW, Dawson R, Shera D. A Multiple Imputation Strategy for Clinical Trials with Truncation of Patient Date. Statistics in Medicine 1995; 14:1913-1925.
- 22. Li X, Mehrotra DV, Barnard J. Analysis of Incomplete Longitudinal Binary Data Using Multiple Imputations. Stat Med. 2006 Jun 30; 25(12):2107-24.
- 23. Lavori PW, Dawson R, Shera D. A multiple imputation strategy for clinical trials with truncation of patient data. Stat Med. 1995; 14:1913-1925.
- 24. Little RJA. Rubin D B. Statistical Analysis with Missing Data. New York: John Wiley &Sons; 1987.
- 25. Rubin DB. Inference and missing data. *Biometrika*. 1976; 63:581-592.
- 26. Little RJA, Schenker N. Handbook of Statistical Methodology-Missing Data. New York: Plenum Press; 1995.
- 27. D'Agostino, R. B., Jr., Rubin, D. B. (2000). Estimating and using propensity scores with partially missing data. Journal of the American Statistical Association 95:749–759
- 28. Yue, L.Q., Lu, N. and Xu, Y., 2014. Designing premarket observational comparative studies using existing data as controls: challenges and opportunities. Journal of biopharmaceutical statistics, 24(5), pp.994-1010.
- 29. Rubin DB. Multiple Imputation for Nonresponse in Surveys. Wiley: New York, 1987.
- 30. Nelson Lu, Yunling Xu, and Lilly Q. Yue (2020) Some Considerations on Design and Analysis Plan on a Nonrandomized Comparative Study Using Propensity Score Methodology for Medical Device Premarket Evaluation, Statistics in Biopharmaceutical Research, 12:2, 155-163, DOI: 10.1080/19466315.2019.1647873

September 04, 2020 

